CLINICAL TRIAL: NCT05480423
Title: A Pilot Study on Application of Online Technology for Mindfulness-based Intervention on Parents of Children With Attention Deficit/Hyperactivity Disorder
Brief Title: Online Mindfulness-based Intervention on Parents of Children With Attention Deficit/Hyperactivity Disorder
Acronym: ADHDparent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ADHDparent
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2022-07

CONDITIONS: Pilot Study
Keywords: ADHD; parent; Mindfulness-based intervention; Online
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online mindfulness-based intervention (Experimental): The online programme lasts for 28 days. Parents will receive the links of daily mini-lectures that introduced basic principles in mindfulness and mindful parenting, audio files of guided mindfulness practice, and exercises that facilitates parents to integrate mindfulness in their daily lives. The total time spent in each session will be around 15 to 20 minutes. Weekly meeting will be arranged with mindfulness instructor and participants.
  Interventions: Behavioral: Mindfulness-based intervention
- Waitlist controlled group (No Intervention): Participants will be offered same intervention three months later

INTERVENTIONS:
Behavioral: Mindfulness-based intervention — 1. Psychoeducation video on mindfulness and mindful parenting. 2. Audio files of mindfulness exercises including mindfulness of breath, body scan, mindful stretching, mindfulness of soles of the feet, befriending exercises. 3. Informal mindfulness exercises by applying mindfulness in daily lives
  Arms: Online mindfulness-based intervention

SUMMARY:
This project apply curriculum of online programme materials and structure for mindful parenting and caregiving. It will include four modules (introductory mindfulness, mindful parenting, applying mindfulness in challenging moments, and advanced exercises for parents of children with special needs). Each module will include short psychoeducation videos and audio mindfulness exercises that can be used in various web-based or application-based platforms. A set of videos and audio exercises will be produced for the core program materials. One study of online mindful parenting program reported a low completion rate below 30%, showing the significance of weekly video or phone contact by professionals in program engagement. Although web-based or application-based mindfulness intervention have become popular, very limited effort has been developed for applying mindfulness in parenting and caregiving using technology. Only two published studies on online mindfulness-based intervention for parents are identified. Objectives of the study are: 1. Investigate the effects of online mindfulness-based intervention for parents of children with Attention Deficit/Hyperactivity Disorder. 2. Validate the protocol of the programme and explore the needs to make refinements of the programme based on the quantitative outcome and qualitative interview analyses

ELIGIBILITY:
Inclusion Criteria:

* parents whose children are between 6 and 18 years old and diagnosed with Attention Deficit/Hyperactivity Disorder
* parents can understand and speak Cantonese Chinese, and
* participants should be the primary caretaker of the children in the last one year

Exclusion Criteria:

* parents who were diagnosed with psychosis, developmental disabilities, or cognitive impairment, which may present difficulties in comprehending the content of the program,
* parents have had prior experience in any 8-week Mindfulness-Based Stress Reduction/Mindfulness-Based Cognitive Therapy or equivalent program.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Parental stress | Change from pre-intervention, to 1-month follow-up, and to 3-month follow-up
  The Parenting Stress Index Short Form (PSI-SF) will be used to measure parental stress (Abidin, 1995; Lam, 1999). A total of 36 items covers three dimensions parental distress, parent-child dysfunctional interaction, and difficult child. Parents will rate the items on a 5-point Likert scale from strongly disagree (1) to strongly agree (5). Total score from 36 to 180. The higher the score, the higher the level of stress.

SECONDARY OUTCOMES:
Parent Anxiety | Change from pre-intervention, to 1-month follow-up, and to 3-month follow-up.
  The anxiety subscale of the Hospital Anxiety and Depression Scale (HADS-A) will be used to measure affective and behavioural symptoms of anxiety (Zigmond & Snaith, 1983). Parents will rate the items on a 4-point Likert scale from 0 to 3, with anchors varying between items (e.g., from "Very much indeed" to "Not at all"). Total score from 0 to 21. The higher the score, the higher the level of anxiety.
Parent depression | Change from pre-intervention, to 1-month follow-up, and to 3-month follow-up
  The 10-item version of the Center for Epidemiologic Studies Depression Scale (CES-D) will be used to measure affective symptoms of depression (Radloff, 1977).Parents will rate the items on a 4-point Likert scale from none of the time (0) to most of the time (3). Total score from 0 to 30. The higher the score, the higher the level of depression.
Family Functioning | Change from pre-intervention, to 1-month follow-up, and to 3-month follow-up.
  The Family Adaptation, Partnership, Growth, Affection, Resolve scale (APGAR) will be used to measure the satisfaction of perceived family functioning (Smilkstein et al., 1982).Parents will rate the items on a 3-point Likert scale from hardly ever (0) to almost always (2). total score from 0 to 10. The higher the score, the higher the level of family functioning.
Parent Quality of Sleep | Change from pre-intervention, to 1-month follow-up, and to 3-month follow-up
  The self-administered version of the Insomnia Severity Index (ISI) will be used to assess sleeping quality (Morin, 1993). The 7-item scale assesses the severity of initial, middle, and late insomnia, distress about sleep difficulties, interference of insomnia with daytime functioning, and notice of sleep problems by others. Parents will rate the items on a 4-point Likert scale from not at all (0) to extremely (2). Total score 0 to 14. The higher the score, the higher the severity of sleep difficulties.
Child Attention Deficit/Hyperactivity Disorder (ADHD) symptomology | Change from pre-intervention, to 1-month follow-up, and to 3-month follow-up.
  The Strengths and Weaknesses of ADHD Symptoms and Normal Behaviors (SWAN) Rating Scale will be used to measure the similarity or differences between a child's attention skills and those of the general population (Swanson et al., 2012). A total of 18 items represents a range of behavioural characteristics. Parents will be asked to compare their child to other same-age children and rate their child on a 7-point Likert scale from far below average (-3) to far above average (3). Total score from -54 to 54. The lower the score, the higher the severity of ADHD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Herman Hay Ming Lo, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lo HHM, Lam J, Zhang ZJ, Cheung M, Chan SKC, Wong EWY, Bogels SM, Chui WH. Effects of an online mindfulness-based program for parents of children with attention deficit/hyperactivity disorder: a pilot, mixed methods study. Front Psychiatry. 2024 Apr 24;15:1376867. doi: 10.3389/fpsyt.2024.1376867. eCollection 2024. PMID 38807691